CLINICAL TRIAL: NCT00981942
Title: An Open Label Clinical Trial of Imatinib Mesylate(Glivec)in Patients With Moderate to Severe Nephrogenic Systemic Fibrosis
Brief Title: Treatment of Patients With Nephrogenic Systemic Fibrosis With Glivec
Acronym: NSF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22505 TRE
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Nephrogenic Systemic Fibrosis
Keywords: Nephrogenic systemic fibrosis; Imatinib mesylate; Glivec; Gleevec
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Imatinib mesylate (Glivec) — 400 mg, one tablet daily for 12 or 24 weeks
  Other Names: Glivec; Gleevec

SUMMARY:
The investigators will study the effect of imatinib mesylate (Glivec) in treatment of moderate to severe nephrogenic systemic fibrosis (NSF).

So far there is no evidence of adequately effective treatment options of NSF. Various treatments have been tried to stop the progressing disease. Corticosteroids, which suppress the early inflammatory stage of the disease, fail to halt disease progression.

Other immunosuppressive agents, photopheresis, and kidney transplantations are reported to be partly beneficial to the patients.

It has not been possible to confirm these findings in further studies because in photopheresis, and kidney transplantation, such effects are generally unreproducible.

DETAILED DESCRIPTION:
NSF is a relatively newly defined fibrosing disease not described before 1997 where the Gadolinium-based contrast agents (GBCAs) were introduced in patients with kidney disease. The association between NSF and GBCA has in many studies shown to be very strong. Until recently, radiologists believed that commercially available GBCAs were safe to use whether the renal function was normal or not. Since the 1980s, >200 million patients have been given these agents. Lately, the occurrence of NSF, a relatively new chronic disorder, has given serious speculations about the safety of these drugs and has questioned their future use. First identified in 1997, but not described until 2000, NSF has been reported only in patients with acute or chronic severe renal insufficiency (with a glomerular filtration rate <30 ml/min/1.73 m2).

Fibrosis in the subcutis means that the skin hardens and loses flexibility. Hard dermal plaque changes often appear on legs, arms and abdomen together with dyspigmentation. As the lesions involve the deep part of the subcutis the muscles are often affected. Involvement of the joints leads to contractures and narrowing of movement. Patients with massive affection of the joints often end up with a zimmer frame or in a wheelchair. The connecting tissue in the inner vital organs may also be affected and NSF can accelerate the death of the patient. The retained gadolinium in lesions of NSF can be found years after administration.

Interestingly, a case report suggests beneficial effects of imatinib mesylate in two patients. Two other independent case reports also show promising results.

Imatinib mesylate inhibits several tyrosine kinases involved in the fibrotic reaction, which is one of the main pathogenetic components of NSF.

ELIGIBILITY:
Inclusion criteria:

1. Age > 18 years
2. Diagnosed with NSF
3. mRodnan skin score => 20 or
4. Rapid progression of the disease defined as a 50% increase in mRodnan skin score in less than 7 weeks or
5. Progression of the fibrosis in the inner organs ex. the heart or the lungs, AND
6. No absolute contraindications to the treatment

Exclusion Criteria:

1. Known sensitivity to Imatinib mesylate or to any of its components
2. Pregnant or lactating woman
3. ALAT > 3 x upper limit of normal
4. Severe congestive heart failure (NYHA Class III or IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are skin fibrosis and joint mobility. | 16 weeks or 28 weeks

SECONDARY OUTCOMES:
The secondary endpoint is and joint mobility. | 16 weeks or 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne B Olesen, MD,PhD, Principal Investigator — Anne Braae Olesen
Locations (2):
- Denmark (2):
  - Department of Dermatology, Aarhus, Aarhus
  - Department of Dermatology, Aarhus

REFERENCES:
- [Background] Kay J, High WA. Imatinib mesylate treatment of nephrogenic systemic fibrosis. Arthritis Rheum. 2008 Aug;58(8):2543-8. doi: 10.1002/art.23696. PMID 18668587